CLINICAL TRIAL: NCT04498949
Title: Transdiagnostic Treatment for University Students at Risk of Emotional Disorders: a Web Based Pilot Randomized Controlled Trial
Brief Title: Transdiagnostic Treatment for Emotional Disorders
Acronym: UP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mohamad hasan yousefi (Other)
Responsible Party: Sponsor-Investigator, Mohamad hasan yousefi, PhD student, Bamyan University
Organization: Bamyan University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Unified Protocol
Record Dates: First submitted 2020-07-16; First posted 2020-08-05 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Depressive Symptoms; Anxiety; Emotional Problem
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exprimental (Experimental): The unified protocol modules are as follows:
  Module 1: Setting the treatment goals and motivation augmentation Module 2: Using psychoeducation to learn the function of emotions and their development Module 3: Mindful (present-focused and non-judgmental) emotional awareness- Core module Module 4: Cognitive flexibility- Core module Module 5: Identifying and countering emotional avoidance behaviors- core module Module 6: Increasing awareness and confronting physical sensations/ interoceptive sensitivity- core module Module 7: Both situational and interoceptive emotion-focused exposures- Core module Module 8: Recognizing accomplishments and looking to the future (relapse prevention)
  Interventions: Behavioral: UP
- Treatment as usual (Active Comparator): Treatment as usual care, Recieve consulting not included unified protocol Recieve supportive cares
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Behavioral: UP — The unified protocol modules are as follows:
  Module 1: Setting the treatment goals and motivation augmentation Module 2: Using psychoeducation to learn the function of emotions and their development Module 3: Mindful (present-focused and non-judgmental) emotional awareness- Core module Module 4: Cognitive flexibility- Core module Module 5: Identifying and countering emotional avoidance behaviors- core module Module 6: Increasing awareness and confronting physical sensations/ interoceptive sensitivity- core module Module 7: Both situational and interoceptive emotion-focused exposures- Core module Module 8: Recognizing accomplishments and looking to the future (relapse prevention)
  Arms: Exprimental
Other: Treatment as usual — Diagnostic test. Psychoeducation Supoortive care
  Other Names: TAU
  Arms: Treatment as usual

SUMMARY:
Background and study aims Depression is more prevalent in younger populations. The age of first onset of depression has become younger, yet many adolescents with depressive symptoms remain untreated. Rates of anxiety and depression are increasing among children and young people.postsecondary education also represents a peak onset period for the occurrence of mental disorders. It is estimated that 12-46% of all university students are affected by mental health disorders in any given year. Who can participate? Afghan students over 18 years old fluent in Persian or Pashto, and access to an internet connection. What does the study involve? Participants will be randomly allocated to receive training in skills and coping strategies which are useful in stressful conditions.

DETAILED DESCRIPTION:
Condition Depressive symptoms, anxiety symptom, emotional problems Interventions Participants in experimental group Receive 12 weeks training according to the guideline below Participants in control Receive treatment as usual, also the experts will respond to their questions. The unified protocol can track its basis from cognitive-behavioral therapy approaches. As in the traditional CBT approaches, the unified protocol has several modules whose base is the emotions . The modules focus on increasing awareness of interaction and the function of the model of emotion components which include thoughts, physical sensations, and behaviors. The final bit of the unified protocol is to change the components to a present moment awareness. The unified protocol is used to treat different emotional disorders unlike the traditional CBT approaches. This is done by targeting the underlying mechanisms that form part of all emotional disorders. The 5 core skills above are delivered to patients through five core modules. Before the key modules, there are 2 modules for introduction and learning about emotions. After the 5 core modules there is a module for treatment progress appraisal and making plans to prevent relapse.

The unified protocol modules are as follows:

Module 1: Setting the treatment goals and motivation augmentation Module 2: Using psychoeducation to learn the function of emotions and their development Module 3: Mindful (present-focused and non-judgmental) emotional awareness- Core module Module 4: Cognitive flexibility- Core module Module 5: Identifying and countering emotional avoidance behaviors- core module Module 6: Increasing awareness and confronting physical sensations/ interoceptive sensitivity- core module Module 7: Both situational and interoceptive emotion-focused exposures- Core module Module 8: Recognizing accomplishments and looking to the future (relapse prevention) Primary outcome measure

At baseline and 12 weeks:

1. Anxiety measured using the Beck Anxiety Inventory (BAI)
2. Depression measured using the Beck Depression Inventory (BDI-II) Secondary outcome measures

At baseline and 12 weeks:

1. Mental health measured using:

   1.1. Overall Anxiety Severity and Impairment Scale (OASIS) 1.2. Overall Depression Severity and Impairment Scale (ODSIS) 1.3. Positive and Negative Affect Scale (PANAS)
2. Quality of life measured using the qolwbref questionnaire) Eligibility Participant inclusion criteria

1. 18 years or older 2. Ability to understand and read Persian or Pashto 3. Access to Internet at home and having an email address 4. Meeting the DSM-IV diagnostic criteria for ED (MDD, DD, MDNOS, PD, A, SAD, GAD, ADNOS, OCD) 5. Providing written, informed consent

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Ability to understand and read Persian or Pashto
* Access to Internet at home and having an email address
* Meeting the DSM-IV diagnostic criteria for ED (MDD, DD, MDNOS, PD, A, SAD, GAD, ADNOS, OCD)

Exclusion Criteria:

* Suffering from a severe mental disorder (schizophrenia, bipolar disorder, and alcohol and/or substance dependence disorder)
* The presence of a high risk of suicide
* other chronic or Medical disease/condition that prevents the participant
* receiving another psychological treatment during the last six month

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 170 (Actual)
Dates: Start 2020-08-15 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Beck anxiety inventory | Baseline
  This is a 21-item self-report questionnaire for the measurement of anxiety symptoms experienced during the past week. Each item is rated from 0 to 3 (i.e. not at all, mildly, moderately, severely), added together to obtain a maximum score of 63. The BAI has demonstrated good to excellent internal consistency in prior validations of the scale (.85-.94), as well as adequate convergent and divergent validity . Cronbach's alpha for the BAI in the present study was excellent
Beck anxiety inventory | 12 weeks after basel8ne
  This is a 21-item self-report questionnaire for the measurement of anxiety symptoms experienced during the past week. Each item is rated from 0 to 3 (i.e. not at all, mildly, moderately, severely), added together to obtain a maximum score of 63. The BAI has demonstrated good to excellent internal consistency in prior validations of the scale (.85-.94), as well as adequate convergent and divergent validity . Cronbach's alpha for the BAI in the present study was excellent
Beck anxiety inventory | Three month follow up
  This is a 21-item self-report questionnaire for the measurement of anxiety symptoms experienced during the past week. Each item is rated from 0 to 3 (i.e. not at all, mildly, moderately, severely), added together to obtain a maximum score of 63. The BAI has demonstrated good to excellent internal consistency in prior validations of the scale (.85-.94), as well as adequate convergent and divergent validity . Cronbach's alpha for the BAI in the present study was excellent
Overall Anxiety Severity and Impairment Scale (OASIS) | 12 weeks after baseline
  he OASIS is a 5-item self-report scale that evaluates the frequency and severity of anxiety symptoms, the functional impairment related to these symptoms (i.e. school, work, home, or social impairment), and behavioral avoidance. Each item instructs respondents to endorse one of five responses that best describes their experiences over the past week. Response items are coded from 0 to 4, added together to obtain a total score ranging from 0 to 20. Previous studies have shown high internal consistency.
Overall Depression Severity and Impairment Scale (ODSIS | Baseline
  .The Overall Depression Severity and Impairment Scale (ODSIS; Bentley et al., 2014) is a 5-item self-report measure that was designed for assessing the frequency and intensity of depression symptoms, the functional impairment related to these depressive symptoms, as well as behavioral avoidance across emotional disorders. Each item of the ODSIS instructs respondents to endorse one of five responses that best describes their experiences over the past week. Response items are coded from 0 to 4 and can be summed to obtain a total score ranging from 0 to 20.
Emotional style questionnaire | baseline
  Emotional style questionnaire consists of 24 items that assess the following dimensions of emotional wellbeing: resilience, outlook; self-awareness, sensitivity to context; social intuition, and attention four item for each sub-scale. Respondents rate the extent to which each item applies to them on a 5-point Likert-type scale from 1 (almost never) to 7 (almost always). Total scores can range from 24 to 168, with higher scores reflecting greater levels of emotional wellbeing.
Emotional style questionnaire | 12 weeks after baseline
  Emotional style questionnaire consists of 24 items that assess the following dimensions of emotional wellbeing: resilience, outlook; self-awareness, sensitivity to context; social intuition, and attention four item for each sub-scale. Respondents rate the extent to which each item applies to them on a 5-point Likert-type scale from 1 (almost never) to 7 (almost always). Total scores can range from 24 to 168, with higher scores reflecting greater levels of emotional wellbeing.
Emotional style questionnaire | Three month follow up
  Emotional style questionnaire consists of 24 items that assess the following dimensions of emotional wellbeing: resilience, outlook; self-awareness, sensitivity to context; social intuition, and attention four item for each sub-scale. Respondents rate the extent to which each item applies to them on a 5-point Likert-type scale from 1 (almost never) to 7 (almost always). Total scores can range from 24 to 168, with higher scores reflecting greater levels of emotional wellbeing.
Difficulties in Emotion Regulation Scale (DERS-16) | Baseline, :
  Difficulties in Emotion Regulation Scale (DERS-16) consists of 16 items that assess the following dimensions of emotion regulation difficulties: nonacceptance of negative emotions (three items), inability to engage in goal-directed behaviors when distressed (three items), difficulties controlling impulsive behaviors when distressed (three items), limited access to emotion regulation strategies perceived as effective (five items), and lack of emotional clarity (two items). As with the original DERS, respondents rate the extent to which each item applies to them on a 5-point Likert-type scale from 1 (almost never) to 5 (almost always). Total scores on the DERS-16 can range from 16 to 80, with higher scores reflecting greater levels of emotion dysregulation.
Difficulties in Emotion Regulation Scale (DERS-16) | 12 weeks after baseline
  Difficulties in Emotion Regulation Scale (DERS-16) consists of 16 items that assess the following dimensions of emotion regulation difficulties: nonacceptance of negative emotions (three items), inability to engage in goal-directed behaviors when distressed (three items), difficulties controlling impulsive behaviors when distressed (three items), limited access to emotion regulation strategies perceived as effective (five items), and lack of emotional clarity (two items). As with the original DERS, respondents rate the extent to which each item applies to them on a 5-point Likert-type scale from 1 (almost never) to 5 (almost always). Total scores on the DERS-16 can range from 16 to 80, with higher scores reflecting greater levels of emotion dysregulation.
Difficulties in Emotion Regulation Scale (DERS-16) | Three month follow up
  Difficulties in Emotion Regulation Scale (DERS-16) consists of 16 items that assess the following dimensions of emotion regulation difficulties: nonacceptance of negative emotions (three items), inability to engage in goal-directed behaviors when distressed (three items), difficulties controlling impulsive behaviors when distressed (three items), limited access to emotion regulation strategies perceived as effective (five items), and lack of emotional clarity (two items). As with the original DERS, respondents rate the extent to which each item applies to them on a 5-point Likert-type scale from 1 (almost never) to 5 (almost always). Total scores on the DERS-16 can range from 16 to 80, with higher scores reflecting greater levels of emotion dysregulation.

SECONDARY OUTCOMES:
The Positive and Negative Affect Schedule or (PANAS) | 12 weeks after baseline
  The Positive and Negative Affect Schedule or (PANAS) is a scale that consists of different words that describe feelings and emotions.The PANAS is designed around 20 items of affect. The scale is comprised of several words that describe different emotions and feelings. (Magyar-Moe, 2009).Scores can range from 10-50 for both the Positive and Negative Affect with the lower scores representing lower levels of Positive/Negative Affect and higher scores representing higher levels of Positive/Negative Affect. (Watson, D., Clark, L. A., & Tellegan, A., 1988).
The Positive and Negative Affect Schedule or (PANAS) | Three months follow up
  The Positive and Negative Affect Schedule or (PANAS) is a scale that consists of different words that describe feelings and emotions.The PANAS is designed around 20 items of affect. The scale is comprised of several words that describe different emotions and feelings. (Magyar-Moe, 2009).Scores can range from 10-50 for both the Positive and Negative Affect with the lower scores representing lower levels of Positive/Negative Affect and higher scores representing higher levels of Positive/Negative Affect. (Watson, D., Clark, L. A., & Tellegan, A., 1988).

CONTACTS AND LOCATIONS:
Locations (1):
- Internet, Bāmyān, Afghanistan

IPD SHARING:
Plan to Share IPD: Yes
Planned publication in a high-impact peer-reviewed journal.
  IPD sharing statement:
  The datasets generated during and/or analysed during the current study are available from the corresponding
Supporting Information: CSR
Time Frame: Between July 2022 to December 2022
Access Criteria: Resonable request via academic email